CLINICAL TRIAL: NCT05600023
Title: The Effectiveness of Single Antibiotic Paste Nitrofurantoin V/S Double Antibiotic Paste in Alleviation of Post-Operative Pain in Adult Patients Symptomatic Irreversible Pulpitis
Brief Title: The Effectiveness of Single Antibiotic Paste Nitrofurantoin Versus Double Antibiotic Paste
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Hira Abbasi, Principal Investigator, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Intracanal medication
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Pain; Symptomatic Irreversible Pulpitis
MeSH Terms: conditions — Pain | interventions — Nitrofurantoin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nitrofurantoin (Experimental)
  Interventions: Drug: Nitrofurantoin
- Double antibiotic paste (Experimental)
  Interventions: Drug: Double Antibiotic
- Control (No Intervention)

INTERVENTIONS:
Drug: Nitrofurantoin — Nitrofurantoin has been found to successfully eradicate gram-negative bacteria such as Enterococcus faecalis that one of the most important bacteria in endodontic lesions
  Arms: Nitrofurantoin
Drug: Double Antibiotic — DAP is a combination of two antibiotics which are ciprofloxacin and metronidazole
  Arms: Double antibiotic paste

SUMMARY:
In our study, we used nitrofurantoin as a root canal medication in patients suffering from symptomatic irreversible pulpitis in alleviating pain compared with double antibiotic paste.

DETAILED DESCRIPTION:
This study aims to compare the efficacy in alleviating pain between intracanal medicaments Nitrofurantoin versus double antibiotic paste.

ELIGIBILITY:
Inclusion Criteria:

* No medical history
* no history of allergy to medications used in root canal treatment
* patients suffering from Symptomatic Irreversible Pulpitis

Exclusion Criteria:

* Patients who were not suitable for conventional root canal treatment
* multirooted teeth

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
To alleviate dental pain | 12 hours upto 72 hours following placement of intracanal medicament
  Dental pain will be measured by using Visual Analogue Scale(VAS) which is an 10-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured

CONTACTS AND LOCATIONS:
Locations (1):
- Hira Danish, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No